CLINICAL TRIAL: NCT00552266
Title: Methylphenidate Treatment of Children and Adolescents Diagnosed With ADHD and Its Influence on Comorbid Trichotillomania
Brief Title: Methylphenidate in ADHD With Trichotillomania
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Geha Mental Health Center (Other)
Collaborators: Clalit Health Services (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pavel1; GMHC2
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: ADHD; Trichotillomania
Keywords: Methylphenidate; Trichotillomania; Attention deficit
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Trichotillomania | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methylphenidate — tablets 10-60 mg/day administered once or twice daily 6 weeks

SUMMARY:
This study will evaluate the safety and effectiveness of methylphenidate in treating attention deficit hyperactivity disorder (ADHD) in children with both ADHD and trichotillomania.

Trichotillomania is an impulse control disorder. There is growing evidences of the involvement of dopaminergic neurotransmission in the pathophysiology of trichotillomania. Reported increase in the prevalence of ADHD among patients with impulse control disorders, such as pathological gambling as well as trichotillomania, may result from the overlapping pathophisiological background. It is hypothesized that in cases of ADHD comorbid with trichotillomania methtylphenidate treatment will exhibit beneficial effects in both the ADHD and the hair pulling.

DETAILED DESCRIPTION:
Thirty children and adolescents aged 6-18 years, diagnosed with ADHD and trichotillomania, will receive MPH monotherapy treatment for a period of 12 weeks, targeting both ADHD and trichotillomania symptoms as rated by the ADHD- rating scale (ADHD-RS) and by the Massachusetts General Hospital Hair Pulling Scale and Clinical Global Impression-Severity (CGI) scale. The rating scales will be assessed at baseline and at the endpoint (after 12 weeks).The side effects will be monitored via weekly spontaneous self reports by each participant. All results will be expressed as mean ±SD. Student's paired t-test and ANOVA test will be used as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Diagnosis of trichotillomania
* DSM-IV diagnosis of ADHD
* Has not taken stimulants or alpha-adrenergic medications for more than 2 weeks prior to entering the study.

Exclusion Criteria:

* History of moderate or severe adverse event, related to MPH
* History of any psychotic disorder
* Current drug abuse, acute psychotic or affective disorder

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Clinicial administered Massachusetts General Hospital Hair Pulling Scale for trichotillomania | First 6 weeks of treatment

SECONDARY OUTCOMES:
Clinicial administered ADHD Rating Scale Clinical Global Impressions (CGI) scale for ADHD severity Weekly spontaneous self report of side effects | Within the first 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Golubchik, M.D., Principal Investigator — Geha Mental Health Center
Locations (1):
- Geha Mental Health Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Golubchik P, Sever J, Weizman A, Zalsman G. Methylphenidate treatment in pediatric patients with attention-deficit/hyperactivity disorder and comorbid trichotillomania: a preliminary report. Clin Neuropharmacol. 2011 May-Jun;34(3):108-10. doi: 10.1097/WNF.0b013e31821f4da9. PMID 21586916